CLINICAL TRIAL: NCT01904799
Title: Cognitive Assessment for Stroke Patients: Reproductibility and Validity Study
Acronym: Casper
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Benaim PHRC N 2012
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Assessment (Other)
  Interventions: Other: Cognitive Assessment test

INTERVENTIONS:
Other: Cognitive Assessment test

SUMMARY:
After a CVA, all of the cognitive functions can be affected and analysed, but the presence of a language disorder may considerably hamper the evaluation of other functions.

The battery of rapid tests to screen for and quantify cognitive disorders, including the MMSE, the MOCA, the R-CAMCOG or the RBANS, are not suitable for aphasic patients because they contain items with a strictly verbal response. Because of this, inexperienced doctors cannot evaluate higher functions (other than language) of aphasics in routine practice. For the same reason, aphasics are regularly excluded from post-cva therapeutic protocols, whether or not the trial bears on the evolution of cognitive functions.

Nonetheless, it is possible to evaluate, at least roughly, all of the cognitive functions without resorting to language.

The investigator have developed , from validated tests and classical clinical manoeuvers, the Cognitive Assessment for Stroke Patients (CASP) :

* for the rapid screening (less than 15 minutes) and quantification of post-cva cognitive disorders (6 functions: language, apraxia, short-term memory, temporal orientation, impaired spatial/visio-construction and executive functions);
* the CASP can be used in most patients, including those with severe disorders of expression and moderate problems with comprehension, The format of these tests has been adapted so that severe disorders of expression (essentially left-hemisphere CVA), and left spatial impairment (right-hemisphere CVA) do not affect the ability to take the test. Its validity in terms of appearance and content were verified in 2011.

ELIGIBILITY:
Inclusion Criteria:

For CVA patients

* patients hospitalised in rehabilitation after a first recent hemispheric CVA (less than 6 weeks) ;
* aged > 18;
* absence of severe disorders of oral comprehension (BDAE aphasia severity score >2 for comprehension);
* whatever the severity of oral expression disorders;
* who have been given clear written and oral information, and after the doctor has verified their ability to understand the protocol.

For " Control " patients (to evaluate divergent validity)

* patients hospitalised in rehabilitation units or geriatrics taking part in this study;
* aged > 18.

Exclusion Criteria:

For CVA patients

* patients who do not speak French;
* cognitive disorders known before the CVA;
* psychotic disorders known before the CVA;
* major visual disorders incompatible with reading, known before the CVA.

For " Control " patients (to evaluate divergent validity)

* patients who do not speak French;
* cognitive disorders known before the CVA;
* psychotic disorders known before the CVA;
* major visual disorders incompatible with reading, known before the CVA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
comprehensive assessment battery of higher functions | baseline
comprehensive assessment battery of higher functions | Evaluation at 3 ±1 days
comprehensive assessment battery of higher functions | Evaluation at 6 ± 2 weeks
test of visual memory | baseline
test of visual memory | Evaluation at 3 ±1 days
test of visual memory | Evaluation at 6 ± 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Benaim C, Wauquiez G, Perennou D, Piscicelli C, Lucas-Pineau B, Bonnin-Koang HY, Vuadens P, Binquet C, Bourredjem A, Devilliers H. Cognitive assessment scale for stroke patients (CASP): A multicentric validation study. Ann Phys Rehabil Med. 2022 May;65(3):101594. doi: 10.1016/j.rehab.2021.101594. Epub 2021 Nov 17. PMID 34687958